CLINICAL TRIAL: NCT05457140
Title: Multiomic Diagnostics in Child and Adolescent Psychosis
Brief Title: Multiomic Diagnostics in Youth With Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Responsible Party: Principal Investigator, Aaron Besterman, Psychiatrist, Clinical Investigator, Rady Pediatric Genomics & Systems Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 801937
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Psychosis
Keywords: Genomic; Pediatric; Rady Children's Hospital
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Enrollees - WGS (Experimental): These participants will be subject to whole genome sequencing and Phage ImmunoPrecipiation sequencing (PhIP-Seq) to identify genetic changes and novel antibodies associated with psychosis.
  Interventions: Genetic: Genetic: Genomic sequencing and molecular diagnostic results, if any.; Diagnostic Test: Phage display ImmunoPrecipiation Sequencing (PhIP-Seq)

INTERVENTIONS:
Genetic: Genetic: Genomic sequencing and molecular diagnostic results, if any. — Genomic sequencing results may be used for diagnosis and treatment of participants.
Diagnostic Test: Phage display ImmunoPrecipiation Sequencing (PhIP-Seq) — Whole Proteome programmable phage display immunoprecipitation sequencing will be used to diagnose known and novel autoantibodies.

SUMMARY:
Rady Children's Institute for Genomic Medicine seeks to understand the genomes and immune systems in 15 children and adolescents who are admitted to Rady Children's Hospital Child and Adolescent Psychiatry Service with psychotic symptoms or schizophrenia. Cutting-edge genome and protein sequencing technology will be used to better understand how immunological and genetic assessments may improve our ability to identify the cause of psychosis and impact care. The investigator also hopes to identify new genetic and/or autoimmune causes of psychosis that may inform new treatment for future patients.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that often starts in late adolescence or early adulthood where individuals experience changes in how they perceive and interact with the world around them (psychosis). These extreme changes in how one perceives and interacts with the world can cause great distress and have a very negative impact on one's life. In most cases, the cause of schizophrenia or psychosis is unknown. However, in a small subset of people who develop schizophrenia or psychosis, their own immune system creates antibodies that attack the brain, which leads to psychosis (autoimmune psychosis). In another subset of patients, there are specific genetic changes that serve as major risk factors for developing psychosis. Identifying autoimmune and genetic factors associated with psychosis with psychosis can inform diagnosis, treatment and prognosis. However, it is still currently unknown how frequently these autoimmune and genetic factors are present in adolescents presenting to the hospital with their first psychotic episode and whether testing for them impacts care.

The investigator proposes a deep analysis of both genomes and immune systems of 15 children and adolescents who are admitted to Rady Children's Hospital Child and Adolescent Psychiatry Service with new psychotic symptoms or schizophrenia. The investigator plans to use cutting-edge genome and protein sequencing technology to better understand how immunological and genetic assessments may improve our ability to identify the cause of psychosis and impact care. The investigator also hopes to identify new genetic and/or autoimmune causes of psychosis that may inform new treatments for future patients.

ELIGIBILITY:
Inclusion Criteria:

Individual in whom one of the following criteria is met:

1. Child/adolescent admitted to the Rady Children's CAPS with symptoms of first break psychosis

   OR
2. Biological parents of child/adolescent enrolled in this study for the purposes of reflex testing. Family members are eligible for participation in this study if they are presumed genetically related to a patient participant.

Exclusion Criteria:

Child/Adolescent patients who do not meet any of the inclusion criteria, or those who:

1. Already received any prior whole genome sequencing or exome sequencing.
2. Unable to approach the family or patient for enrollment.
3. Unable to obtain informed consent.
4. Family members are ineligible for participation in this study if:

   1. They are known to not be genetically related to the child/adolescent patient participant
   2. They are a member of a protected research population

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of brain reactive autoantibodies | 2 years
  Diagnostic rate of brain reactive autoantibodies via genomic and whole human proteome programmable phage display immunoprecipitation sequencing (PhIP-Seq)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Besterman, MD, Principal Investigator — Rady Pediatric Genomics & Systems Medicine Institute
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States